CLINICAL TRIAL: NCT04097574
Title: Phase II Study of NPO-13 in Patients Undergoing Colonoscopy
Brief Title: Study of NPO-13 During Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NPO-13-01/ED-01
Record Dates: First submitted 2019-08-20; First posted 2019-09-20 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Bowel Disease
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NPO-13 0.8% (Active Comparator): Low dose
  Interventions: Drug: NPO-13: l-menthol
- NPO-13 1.6% (Active Comparator): High dose
  Interventions: Drug: NPO-13: l-menthol
- NPO-13 0% (Placebo Comparator): Placebo
  Interventions: Drug: NPO-13: l-menthol

INTERVENTIONS:
Drug: NPO-13: l-menthol — 20 mL/site

SUMMARY:
This study will investigate the safety, efficacy and dose-response of NPO-13 in subjects with moderate to severe colonic spasm during colonoscopy. An intraluminal spraying of NPO-13 dosed up to twice into ascending or sigmoid colon. The colonic spasm will be assessed by an independent committee using recorded video images. The study consists of a screening visit window, 1-day treatment phase and 1-week follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are between 20 and 85 years at the time of consent
2. Patients who need colonoscopy

Exclusion Criteria:

1. Patients with a history of abdominal surgical treatment (including the laparoscopic surgery) including the gynecology operation
2. Patients with contraindication to colonoscopy including the paralytic ileus
3. Patients with a history of shock or hypersensitivity to l-menthol or peppermint oil (mint oil)
4. Patient with contraindication to bowel cleansing preparation
5. Patient with contraindication to pain medicine and sedative medicine
6. Patient with contraindication to butylscopolamine bromide and glucagon
7. Patients on cancer treatment (chemotherapy or radiotherapy)
8. Patient with active inflammatory bowel disease or infectious enteritis
9. Patients who need sedative in colonoscopy
10. Patients who receives a therapeutic colonoscopy
11. Pregnant or lactating women, women of childbearing potential, or women who plan to become pregnant during the study
12. Patients who have received other investigational drugs within four months before consent or who are participating in other clinical studies
13. Patients otherwise ineligible for participation in the study in the investigator's or coinvestigator's opinion

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Proportion of No or Mild colonic spasm at the all sites of NPO-13 treatment | 3 minutes
  The primary endpoint will be evaluated by third-party organization, using a four-grade scale: 1, No; 2, Mild; 3, Moderate; 4, Severe.

SECONDARY OUTCOMES:
Proportion of No or Mild colonic spasm at the each site of NPO-13 treatment | 3 minutes
  The secondary endpoint will be evaluated by third-party organization, using a four-grade scale: 1, No; 2, Mild; 3, Moderate; 4, Severe.
Change in colonic spasm before and after treatment of NPO-13 treatment | 3 minutes
  The evaluated colonic spasm grades will be converted into a numeric score, and difference between paired mean scores (before and after application, or 0.8% NPO-13, 1.6% NPO-13 and placebo) will be calculated.
Time to effect | 3 minutes
  The onset of anti-spasmodic effect is the interval from the spray to the disappearance of the spasm.
Difficulty of endoscopic observation | 3 minutes
  The proportion of subjects in whom intracolonic examination will be evaluated by the investigator to be "Very easy" or "Easy"., using a four-grade scale: 1, Very easy; 2, Easy; 3, Difficult; 4, Hard.
Adverse events and Adverse drug reactions | 7 ± 3 days
  The subjects will be observed for 7 days after colonoscopy, and all adverse events and adverse drug reactions will be recorded and compared with the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Hisatsugu Asada, Study Chair — Nihon Pharmaceutical Co., Ltd
Locations (13):
- Japan (13):
  - NPO-13 Trial Site 11, Kitakyushu, Fukuoka
  - NPO-13 Trial Site 12, Kurume, Fukuoka
  - NPO-13 Trial Site 2, Maebashi, Gunma
  - NPO-13 Trial Site 5, Yokohama, Kanagawa
  - NPO-13 Trial Site 6, Yokohama, Kanagawa
  - NPO-13 Trial Site 1, Shimotsuke, Tochigi
  - NPO-13 Trial Site 4, Minato, Tokyo
  - NPO-13 Trial Site 3, Shinjuku, Tokyo
  - NPO-13 Trial Site 9, Hiroshima
  - NPO-13 Trial Site 13, Kagoshima
  - NPO-13 Trial Site 10, Kochi
  - NPO-13 Trial Site 7, Osaka
  - NPO-13 Trial Site 8, Osaka

IPD SHARING:
Plan to Share IPD: No